CLINICAL TRIAL: NCT06192056
Title: Feasibility and Preliminary Efficacy of Web-Based Self-Help Program on Repetitive Negative Thinking for College Students: A Randomized Pilot Study
Brief Title: Feasibility and Preliminary Efficacy of a Web-Based Self-Help Program for College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CanSagligi Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSV202302
Record Dates: First submitted 2023-12-07; First posted 2024-01-05 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Repetitive Negative Thinking
Keywords: Acceptance and Commitment Therapy; Rumination
MeSH Terms: conditions — Rumination Syndrome

STUDY DESIGN:
Intervention Model Description: Intervention group vs waitlist group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The RNT-focused web based self-help program will be given to the intervention group.
  Interventions: Behavioral: RNT Focused Web- Based Self-Help Program
- Waitlist group (No Intervention): Waitlist group will be given only pre and post test measures at the same time with the intervention group.

INTERVENTIONS:
Behavioral: RNT Focused Web- Based Self-Help Program — This 10 day long intervention contains psychoeducational contents, experimental exercises, monitoring behavior and committed action strategies. Each step of the intervention aims to develop a specific psychological flexibility skill like cognitive defusion etc.
  Arms: Intervention group

SUMMARY:
The goal of this pilot study is to test the feasibility and preliminary efficacy of the repetitive negative thinking (RNT) focused web-based self-help program in college students. The main questions it aims to answer are:

* Does the program work without any help of a clinician?
* Does the program have any reducing effect on the participants' RNT, depression, anxiety, stress and cognitive fusion scores? - Does the program help participants to improve their psychological flexibility and committed actions? Participants will be administered a set of questionnaires before and after completing the 10-day long web-based self-help program, provided on a daily basis. Researchers will compare the intervention group with a waitlist control group to assess for any potential placebo effect.

DETAILED DESCRIPTION:
After obtaining informed consent, all participants will receive a set of questionnaires for baseline measurement. Participants will be randomized into two groups using block randomization: one as the intervention group and the other as the control group (waitlist condition). This method helps ensure an equal distribution of participants with similar characteristics in both groups, minimizing potential biases and increasing the validity of the study.

ELIGIBILITY:
Inclusion Criteria:

* having internet connection and a working smart phone or computer

Exclusion Criteria:

* having thoughts of self-harm or suicide,
* diagnosed with psychotic disorder,
* substance abuse
* currently receiving psychological help

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Perseverative Thinking Questionnaire (PTQ) Scores | Baseline and Week 2
  The PTQ is a validated self-report instrument assessed content-independent trait-based RNT. It consists of 15 items that rated on the score of 0 (never) to 4 (almost always). The reliability and validity of the Turkish version of the scale is checked and it found suitable for Turkish population. Change (Post-intervention score- Baseline score)

SECONDARY OUTCOMES:
Improvement in Cognitive Fusion Questionnaire (CFQ) Scores | Baseline and Week 2
  Improvement is defined as a significant reduce in participants' CFQ scores. Turkish version of CFQ is a 7-item questionnaire assessed on 7-point Likert-type scale (1: "Never true"; 7: "Always true"). The validity and reliability study for Turkish version of the CFQ was conducted.
Enhancement in Psychological Flexibility measured by Acceptance and Action Questionnaire (AAQ-II) | Baseline and Week 2
  The AAQ-II is a validated self-report instrument designed to measure psychological inflexibility. Higher scores on the AAQ-II indicate greater psychological inflexibility. The 7-item questionnaire has been found to be reliable and valid in Turkish.
Change from Baseline in Depression Anxiety Stress Scale-21 (DASS-21) Scores | Baseline and Week 2
  The DASS-21 consists of three subscales, each with 7 items rated on a scale of 0 (never) to 3 (always). The scale assesses depression, anxiety, and stress levels in the past week. The Turkish version of the scale has been found to be reliable and valid. Change (Post-intervention score- Baseline score)
Increase in Committed Actions | Baseline and Week 2
  The change in participants' committed actions in life is measured by the Valuing Questionnaire (VQ). The questionnaire comprises 10 items rated on a 7-point Likert scale (0=Not at all true; 6=Completely true). A higher score on the scale indicates that individuals are behaving in a manner consistent with their values. Change (Post-intervention score- Baseline score)
System Usability Assessment | Week 2
  The Turkish version of the System Usability Scale (SUS) will be administered at the conclusion of the 10-day web-based self-help program to assess the understandability and applicability of the program for participants. The SUS is a 10-item standardized questionnaire that offers a subjective assessment of usability. Participants rate the items on a scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree).

CONTACTS AND LOCATIONS:
Overall Officials: Fatih K Yavuz, Principal Investigator — İstanbul Medipol University
Locations (1):
- CanSagligi Foundation, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data would be available upon request.